CLINICAL TRIAL: NCT00862797
Title: Pressure Course in the Tube Cuff During Swallowing
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. med. Daniel Steinmann, University Medical Center Freiburg
Other Study IDs: 273/07
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-03

CONDITIONS: Anesthesia; Intensive Care
Keywords: endotracheal tube; swallowing; aspiration; cuff pressure; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- endotracheal tube: Patients intubated with cuffed endotracheal tubes
  Interventions: Other: pressure measurement during swallowing

INTERVENTIONS:
Other: pressure measurement during swallowing — measurement of endotracheal tube cuff pressure during swallowing while recovering from anaesthesia

SUMMARY:
Leakage of fluid from the subglottic space to the lungs occurs along the longitudinal folds within the wall of endotracheal tube (ETT) cuffs. In this project the researchers investigate the possible effect of swallowing on the pressure course in the ETT cuff.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* general anaesthesia or intensive care medicine treatment

Exclusion Criteria:

* refusal of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recovering from general anaesthesia or intensive care patients both intubated with cuffed endotracheal tubes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinmann, MD, Principal Investigator — University Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany